CLINICAL TRIAL: NCT02626923
Title: Observational Study of the Safety and Efficacy of Nucleoside Reverse Transcriptase Inhibitor Backbones With Maraviroc (MVC) and Epzicom (ABC/3TC) Once-Daily in Antiretroviral Therapy-Naive Patients and First-Switch Subjects
Brief Title: Study of Maraviroc (MVC) and Epzicom (ABC/3TC) Once-Daily in ART-Naive & First Switch Patients
Status: Completed | Type: Observational
Sponsor: Nicholaos C Bellos, MD (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Nicholaos C Bellos, MD, MD, Southwest Infectious Disease Clinical Research, Inc.
Organization: Southwest Infectious Disease Clinical Research, Inc. (Other)
Other Study IDs: 759-TBC
Record Dates: First submitted 2015-12-07; First posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Drug-induced Hypotension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients on once daily Maraviroc: Maraviroc tablet 600 mg once daily 48 weeks

SUMMARY:
Hypotension does not occur with Maraviroc at a dose of 600 mg/day

DETAILED DESCRIPTION:
A qualitative description of orthostatic hypotension in patients receiving once daily Maraviroc at 600 mg with Epzicom measured by a validated questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Epzicom Maraviroc once daily dosing

Exclusion Criteria:

* Maraviroc with any other back bone

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV impacted individual on therapy with once daily Maraviroc
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2012-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Hypotension related to once daily Maraviroc dosing | 48 Weeks
  Blood pressure lowering secondary to Maraviroc 600 mg once daily dosing

CONTACTS AND LOCATIONS:
Overall Officials: Nicholaos C Bellos, MD, Study Chair — Southwest Infectious Disease, PA